CLINICAL TRIAL: NCT02681900
Title: Exploring Whether Experimentally Manipulated Self-affirmation Promotes Reduced Alcohol Consumption in Response to Narrative Health Information
Brief Title: Exploring Whether Self-affirmation Promotes Reduced Alcohol Consumption in Response to Narrative Health Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sussex (Other)
Collaborators: Economic and Social Research Council, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ER/KJF25/4
Record Dates: First submitted 2016-02-02; First posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-affirmation (Experimental): Participants in the self-affirmation arm write about their most important value, reasons why is important and an example of when they enacted that value. This is the Self-affirmation manipulation task as described in the intervention.
  Interventions: Behavioral: Self-affirmation manipulation task
- Control (Active Comparator): Participants in this arm complete a control equivalent of the self-affirmation task, where they write about their least important value, reasons why is may be important to someone else and an example of when another person may have enacted that value. This is the Control task as described in the intervention.
  Interventions: Behavioral: Control task

INTERVENTIONS:
Behavioral: Self-affirmation manipulation task — Participants in the self-affirmation condition indicate their most important value, give three examples of why this value is important to them and one example of something they had done to demonstrate its importance.
  Arms: Self-affirmation
Behavioral: Control task — People in the control condition indicate their least important value, three examples of why that value could be important to someone else, and describe something that person could do to show its importance.
  Arms: Control

SUMMARY:
This study tests the effects of a self-affirmation manipulation on (i) acceptance of a health message detailing the risks of alcohol consumption, (ii) engagement with the health message and (iii) alcohol consumption at 7-day follow-up. Half of the participants complete a self-affirmation manipulation, where they reflect on their most important values, whereas the other half complete a control equivalent, where they reflect on their least important values. Immediately post-intervention, all participants then receive information about the risks of alcohol consumption and complete measures of message acceptance and engagement with the materials. Seven days after intervention, participants self-report their alcohol consumption in the previous 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Drinkers

Exclusion Criteria:

* Male
* Non-drinkers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption 7 days after intervention | 7 days after intervention
  Seven days after the intervention, participants are contacted and asked to report their alcohol consumption over the previous 7-day period via self-report items. Participants report the type of alcohol (e.g., beer, spirit), type of container (e.g., small glass, pint, single measure) and the number of each type of drink they had consumed on each day over the previous 7 days using the adapted version (Armitage, Harris, & Arden, 2011) of the timeline fallback technique (Sobell & Sobell, 1992). The total number of units consumed by each participant was then calculated using the UK NHS alcohol unit calculator (NHS Choices, 2013: www.nhs.uk/tools/pages/alcohol-unit-calculator.aspx).

SECONDARY OUTCOMES:
Effect of intervention on acceptance of health information | Immediately after intervention
  Measures to assess whether the intervention affected the extent to which people accepted information about the risks of alcohol consumption were taken immediately after the intervention via self-report items. Acceptance items included personal relevance, negative affect, attitudes, anticipated regret and intentions. Responses to items were given on 7-point scales with relevant anchors (e.g. strongly disagree [1] to strongly agree [7]). A mean score was calculated for each participant on each measure, with higher scores indicating greater levels of that construct.
Effect of intervention on engagement with health information | Immediately after intervention
  Measures to assess whether the intervention affected the extent to which people engaged with the information were taken immediately after the intervention via self-report items. Engagement items included perspective taking, attention, emotion and visualization. Responses to items were given on 7-point scales with relevant anchors (e.g. strongly disagree [1] to strongly agree [7]). A mean score was calculated for each participant on each measure, with higher scores indicating greater levels of that construct.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry J Fox, MSc, Principal Investigator — University of Sussex
Locations (1):
- University of Sussex, Falmer, Brighton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fox KJ, Harris PR, Jessop DC. Experimentally Manipulated Self-Affirmation Promotes Reduced Alcohol Consumption in Response to Narrative Information. Ann Behav Med. 2017 Dec;51(6):931-935. doi: 10.1007/s12160-017-9912-2. PMID 28484982